CLINICAL TRIAL: NCT02192190
Title: A Phase 2, Randomized, Double-Blind, Placebo and Active-Controlled Trial of LY2951742 in Patients With Mild to Moderate Osteoarthritis Pain of the Knee
Brief Title: A Study of LY2951742 in Participants With Mild to Moderate Osteoarthritis Knee Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim assessment: Lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15515; I5Q-MC-CGAF (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — galcanezumab; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Placebo capsule orally, once daily for approximately 16 weeks. Placebo subcutaneous (SC) once every 4 weeks for 16 weeks (Treatment period = 16 weeks).
  Interventions: Other: Placebo- oral; Other: Placebo - SC
- Celecoxib + Placebo (Active Comparator): Celecoxib 200 milligram (mg) capsule orally once daily for approximately 16 weeks. Placebo SC once every 4 weeks for 16 weeks (Treatment period = 16 weeks).
  Interventions: Other: Placebo - SC; Drug: Celecoxib
- LY2951742 5 mg + Placebo (Experimental): Placebo capsule orally, once daily for approximately 16 weeks. SC injections of 5 mg LY2951742 once every 4 weeks for 8 weeks followed by placebo SC once every 4 weeks for 8 weeks (Treatment period = 16 weeks).
  Interventions: Drug: LY2951742; Other: Placebo- oral; Other: Placebo - SC
- LY2951742 50 mg + Placebo (Experimental): Placebo capsule orally, once daily for approximately 16 weeks. SC injections of 50 mg LY2951742 once every 4 weeks for 8 weeks followed by placebo SC once every 4 weeks for 8 weeks (Treatment period = 16 weeks).
  Interventions: Drug: LY2951742; Other: Placebo- oral; Other: Placebo - SC
- LY2951742 120 mg + Placebo (Experimental): Placebo capsule orally, once daily for approximately 16 weeks. SC injections of 120 mg LY2951742 once every 4 weeks for 8 weeks followed by placebo SC once every 4 weeks for 8 weeks (Treatment period = 16 weeks).
  Interventions: Drug: LY2951742; Other: Placebo- oral; Other: Placebo - SC
- LY2951742 300 mg + Placebo (Experimental): Placebo capsule orally, once daily for 16 weeks. SC injections of 300 mg LY2951742 once every 4 weeks for 8 weeks followed by placebo SC once every 4 weeks for 8 weeks (Treatment period = 16 weeks).
  Interventions: Drug: LY2951742; Other: Placebo- oral; Other: Placebo - SC

INTERVENTIONS:
Drug: LY2951742 — Administered subcutaneously (SC)
  Arms: LY2951742 120 mg + Placebo; LY2951742 300 mg + Placebo; LY2951742 5 mg + Placebo; LY2951742 50 mg + Placebo
Other: Placebo- oral — Administered orally
  Arms: LY2951742 120 mg + Placebo; LY2951742 300 mg + Placebo; LY2951742 5 mg + Placebo; LY2951742 50 mg + Placebo; Placebo
Other: Placebo - SC — Administered SC
Drug: Celecoxib — Administered orally
  Arms: Celecoxib + Placebo

SUMMARY:
The main purpose of this study is to test if LY2951742 relieves mild to moderate knee pain. The study drugs will be given as an injection under the skin and as an oral capsule. The study will last about 28 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have osteoarthritis (OA) of the knee joint based on American College of Rheumatology (ACR) criteria and confirmed with X-rays and ACR functional class of I to III
* Have been on stable dose of prescription Nonsteroidal Anti-Inflammatory Drugs (NSAIDS), celecoxib, tramadol, or acetaminophen of at least 2000 mg per day for at least 20 days in the past month
* Willing to stop all analgesics for OA pain during the study
* Experienced pain while walking in the target knee of 50-90 mm inclusive on 0-100 Visual Analog Scale (VAS) with an increase in pain while walking of at least 10 mm following washout of current Osteoarthritis pain medications at screening

Exclusion Criteria:

* Allergic to LY2951742, celecoxib, other NSAIDS, including aspirin, and similar drugs
* Arthritis of the knee from other causes
* Uncontrolled hypertension
* Have OA pain that requires treatment with potent opioids, systemic corticosteroids, intra-articular injections, duloxetine, or venlafaxine
* Moderate to severe renal impairment
* Pregnant or lactating

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- United States (38):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Dream Team Clinical Research, Anaheim, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Empire Clinical Research, Upland, California
  - Diablo Clinical Research, Walnut Creek, California
  - iM Research, West Covina, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Avail Clinical Research LLC, DeLand, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Community Research Foundation Inc, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - M&M Medical Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, Orlando, Florida
  - United Osteoporosis Center, Gainesville, Georgia
  - Drug Studies America, Marietta, Georgia
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - ActivMed Practices & Research, Inc, Methuen, Massachusetts
  - The Center for Clinical Trials, Inc., Biloxi, Mississippi
  - Arthritis, Rheumatic & Back Disease Associates, Voorhees Township, New Jersey
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Drug Trials of America, Hartsdale, New York
  - Medex Healthcare Research, Inc., New York, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - PharmQuest, Greensboro, North Carolina
  - Family Practice Center of Wooster, Wooster, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Greater Providence Clinical Research, LLC, Warwick, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - PCPMG Clinical Research Unit, Greenville, South Carolina
  - Accurate Clinical Research, Nassau Bay, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Health Research of Hampton Roads Inc, Newport News, Virginia
  - National Clinical Research - Norfolk Inc, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jin Y, Smith C, Monteith D, Brown R, Camporeale A, McNearney TA, Deeg MA, Raddad E, Xiao N, de la Pena A, Kivitz AJ, Schnitzer TJ. CGRP blockade by galcanezumab was not associated with reductions in signs and symptoms of knee osteoarthritis in a randomized clinical trial. Osteoarthritis Cartilage. 2018 Dec;26(12):1609-1618. doi: 10.1016/j.joca.2018.08.019. Epub 2018 Sep 18. PMID 30240937

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo capsule orally, once daily for 16 weeks. Placebo subcutaneous (SC) once every 4 weeks for 16 weeks.
- Celecoxib: Celecoxib 200 milligram (mg) capsule orally once daily for 16 weeks. Placebo SC once every 4 weeks for 16 weeks.
- LY2951742 5 mg + Placebo: Placebo capsule orally, once daily for 16 weeks. SC dose of 5 mg LY2951742 once every 4 weeks for 16 weeks.
- LY2951742 50 mg + Placebo: Placebo capsule orally, once daily for 16 weeks. SC injection of 50 mg LY2951742 once every 4 weeks for 16 weeks.
- LY2951742 120 mg + Placebo: Placebo capsule orally, once daily for 16 weeks. SC injections of 120 mg LY2951742 once every 4 weeks for 16 weeks.
- LY2951742 300 mg + Placebo: Placebo capsule orally, once daily for 16 weeks. SC injections of 300 mg LY2951742 once every 4 weeks for 16 weeks.
Period: Overall Study
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Started | 76 | 39 | 38 | 38 | 39 | 38
Received at Least 1 Dose of Study Drug | 76 | 39 | 38 | 38 | 38 | 37
Completed | 22 | 10 | 13 | 12 | 9 | 9
Not Completed | 54 | 29 | 25 | 26 | 30 | 29
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 3 | 2 | 1 | 4 | 3
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Terminated by Sponsor | 43 | 23 | 20 | 23 | 21 | 23
Not completed — Withdrawal by Subject | 4 | 1 | 2 | 1 | 5 | 3
Not completed — Could not Keep Visit Schedule | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Positive Drug Screen | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Inadequate Pain Relief | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo | Total
Number analyzed (Participants) | 76 | 39 | 38 | 38 | 38 | 37 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (7.94) | 60.8 (9.86) | 58.0 (9.60) | 56.7 (7.95) | 58 (9.29) | 56.4 (9.38) | 58.2 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 24 | 23 | 22 | 23 | 19 | 164
  Male | 23 | 15 | 15 | 16 | 15 | 18 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 21 | 17 | 19 | 19 | 17 | 135
  Not Hispanic or Latino | 34 | 18 | 21 | 19 | 18 | 20 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 7 | 11 | 13 | 12 | 13 | 75
  White | 54 | 31 | 25 | 25 | 23 | 23 | 181
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 8 Weeks in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale
Description: The 24-question WOMAC Osteoarthritis Index assesses osteoarthritis (OA) symptoms using pain (5 questions), stiffness (2 questions) and physical function (17 questions) subscales. The WOMAC pain subscale was calculated for each participant at each time point for analysis as the mean score (range 0-100 millimeter [mm] VAS; 0=very good and 100=very poor) of all 5 questions related to pain. Bayesian posterior adjusted mean was calculated using a Bayesian Normal Dynamic Linear Model (NDLM) dose response model with baseline and pooled investigator site included as baseline covariates.
Time Frame: Baseline, 8 Weeks
Population: Full Analysis Set (FAS) is the number of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose baseline efficacy assessment. N = participants in the full analysis set with an evaluable WOMAC assessment at weeks 2, 4, 6 or 8. The 95% Crl (Credible Interval) is reported, not confidence interval (CI).
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Number analyzed (Participants) | 65 | 32 | 31 | 31 | 30 | 30
mm | -19.2 [-24.7 to -13.4] | -31.3 [-40.1 to -22.5] | -16.4 [-23.9 to -8.6] | -24.2 [-31.0 to -17.2] | -21.8 [-29.3 to -14.2] | -17.7 [-25.2 to -10.0]

2. Secondary Outcome: Change From Baseline to 8 Weeks in the WOMAC Physical Function Subscale
Description: The 24-question WOMAC Osteoarthritis Index assesses osteoarthritis symptoms using pain (5 questions), stiffness (2 questions) and physical function (17 questions) subscales. The WOMAC Osteoarthritis Index version 3.1 was administered according to the study schedule. The WOMAC physical function subscale was calculated for each participant at each time point for analysis as the mean score (range 0-100 mm VAS; 0=very good and 100=very poor) of all 17 questions related to physical function. Least Square Mean (LSM) was calculated using a mixed-effects model repeated measures (MMRM) approach with treatment, visit and the interaction of treatment and visit were fitted as fixed effects in the model and baseline and pooled investigator site as baseline covariates.
Time Frame: Baseline, 8 Weeks
Population: FAS: Randomized participants who received at least 1 dose of study drug and had at least 1 post-dose baseline efficacy assessment. N = participants in the full analysis set with an evaluable WOMAC assessment at weeks 2, 4, 6 or 8.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Number analyzed (Participants) | 65 | 32 | 31 | 31 | 30 | 30
mm | -16.5 [-22.3 to -10.8] | -30.6 [-38.8 to -22.4] | -15.4 [-23.7 to -7.12] | -23.5 [-31.4 to -15.6] | -19.5 [-28.2 to -10.9] | -18.4 [-26.8 to -9.9]

3. Secondary Outcome: Change in Baseline to 8 Weeks in Patient's Global Assessment of Osteoarthritis
Description: The PGA is a patient-rated instrument that measures their assessment of overall OA symptoms. It is based on the participant's response to the question "Considering all the ways your osteoarthritis affects you, how are you doing today?" using a 100 mm VAS (0=very good and 100=very poor). LSM mean was calculated using a mixed-effects model repeated measures (MMRM) approach with treatment, visit and the interaction of treatment and visit were fitted as fixed effects in the model and baseline and pooled investigator site as baseline covariates.
Time Frame: Baseline, 8 Weeks
Population: FAS: Randomized participants who received at least 1 dose of study drug and had at least 1 post-dose baseline efficacy assessment. N = participants in the full analysis set with an evaluable PGA assessment at weeks 2, 4, 6 or 8.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Number analyzed (Participants) | 62 | 31 | 29 | 30 | 28 | 28
mm | -22.5 [-28.8 to -16.2] | -36.7 [-45.7 to -27.6] | -18.5 [-27.9 to -9.1] | -19.4 [-28.0 to -10.8] | -21.2 [-31.2 to -11.1] | -20.4 [-30.0 to -10.9]

4. Secondary Outcome: Number of Participants With a Response Rate Measured by the Outcome Measures for Rheumatology Committee and Osteoarthritis Research Society International Standing Committee for Clinical Trials Response Criteria Initiative (OMERACT-OARSI)
Description: The responders according to OMERACT-OARSI criteria: participants with at least 50 % improvement in pain or in function scores, along with absolute improvement of 20 mm, were considered responders. Alternatively, participants were considered responders if they showed at least 20% improvement and absolute improvement of 10 mm in at least two of the following scores: pain, function and Patients Global Assessment (PGA) scores.
Time Frame: 8 Weeks
Population: FAS: Randomized participants who received at least 1 dose of study drug and had at least one post-dose efficacy assessment. N= participants analyzed in the full analysis set with an evaluable response rate at week 8.
Measure: Number; unit: participants
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Number analyzed (Participants) | 41 | 20 | 29 | 22 | 16 | 19
participants | 21 | 14 | 7 | 15 | 10 | 10

5. Secondary Outcome: Change From Baseline to 8 Weeks in the WOMAC Stiffness Subscale
Description: The 24-question WOMAC Osteoarthritis Index assesses osteoarthritis symptoms using pain (5 questions), stiffness (2 questions) and physical function (17 questions) subscales. The WOMAC stiffness subscale will be calculated for each participant at each time point for analysis as the mean score (range 0-100 mm VAS; 0=very good and 100=very poor) of 2 questions related to stiffness. LSM mean was calculated using a mixed-effects model repeated measures (MMRM) approach with treatment, visit and the interaction of treatment and visit were fitted as fixed effects in the model and baseline and pooled investigator site as baseline covariates. LSM mean was calculated using a mixed-effects model repeated measures (MMRM) approach with treatment, visit and the interaction of treatment and visit were fitted as fixed effects in the model and baseline and pooled investigator site as baseline covariates.
Time Frame: Baseline, 8 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Number analyzed (Participants) | 65 | 32 | 31 | 31 | 30 | 30
mm | -18.5 [-24.6 to -12.4] | -31.4 [-40.1 to -22.7] | -15.1 [-24.0 to -6.3] | -23.7 [-32.1 to -15.4] | -21.3 [-30.7 to -12.0] | -17.3 [-26.2 to -8.3]

6. Secondary Outcome: Change From Baseline to 8 Weeks in the WOMAC Total Score
Description: The 24-question WOMAC Osteoarthritis Index assesses osteoarthritis symptoms using pain (5 questions), stiffness (2 questions) and physical function (17 questions) subscales.The WOMAC total score was calculated for each participant at each time point for analysis as the mean score (range 0-100 mm VAS; 0=very good and 100=very poor) of 24 questions. LSM mean was calculated using a mixed-effects model repeated measures (MMRM) approach with treatment, visit and the interaction of treatment and visit were fitted as fixed effects in the model and baseline and pooled investigator site as baseline covariates. LSM mean was calculated using a mixed-effects model repeated measures (MMRM) approach with treatment, visit and the interaction of treatment and visit were fitted as fixed effects in the model and baseline and pooled investigator site as baseline covariates.
Time Frame: Baseline, 8 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Number analyzed (Participants) | 65 | 32 | 31 | 31 | 30 | 30
mm | -17.0 [-22.7 to -11.4] | -31.1 [-39.2 to -23.0] | -15.6 [-23.8 to -7.47] | -23.7 [-31.5 to -15.9] | -20.0 [-28.5 to -11.5] | -18.4 [-26.7 to -10.1]

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Celecoxib | LY2951742 5 mg + Placebo | LY2951742 50 mg + Placebo | LY2951742 120 mg + Placebo | LY2951742 300 mg + Placebo
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/39 | 0/38 | 0/38 | 0/38 | 1/37
Other Adverse Events (participants affected / at risk) | 27/76 | 13/39 | 8/38 | 8/38 | 13/38 | 9/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Celecoxib (N=39) | LY2951742 5 mg + Placebo (N=38) | LY2951742 50 mg + Placebo (N=38) | LY2951742 120 mg + Placebo (N=38) | LY2951742 300 mg + Placebo (N=37)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Celecoxib (N=39) | LY2951742 5 mg + Placebo (N=38) | LY2951742 50 mg + Placebo (N=38) | LY2951742 120 mg + Placebo (N=38) | LY2951742 300 mg + Placebo (N=37)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Computerised tomogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 1 (3) | 0 (0) | 1 (1) | 1 (3) | 3 (3)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days